CLINICAL TRIAL: NCT00963105
Title: A Phase 2, Multi-Center, Randomized, Double-Blinded, Parallel Group Study of the Safety and Efficacy of Different Lenalidomide (REVLIMID®) Dose Regimens in Subjects With Relapsed or Refractory B-Cell Chronic Lymphocytic Leukemia
Brief Title: Study of Lenalidomide to Evaluate Safety and Efficacy in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-5013-CLL-009; 2009-009836-54 (EudraCT Number)
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Relapsed or Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lenalidomide 5 mg (Experimental): Participants received a starting dose of 5 mg lenalidomide orally once a day. Lenalidomide dose was escalated by 5 mg in a step-wise manner every 28 days up to a maximum dose of 25 mg daily based on tolerability.
  Participants continued receiving study drug until disease progression or unacceptable toxicity, unless they withdrew consent or had other reasons to discontinue from study drug
  Interventions: Drug: lenalidomide
- Lenalidomide 10 mg (Experimental): Participants received a starting dose of 10 mg lenalidomide orally once a day. Lenalidomide dose was escalated by 5 mg in a step-wise manner every 28 days up to a maximum dose of 25 mg daily based on tolerability.
  Participants continued receiving study drug until disease progression or unacceptable toxicity, unless they withdrew consent or had other reasons to discontinue from study drug
  Interventions: Drug: lenalidomide
- Lenalidomide 15 mg (Experimental): Participants received a starting dose of 15 mg lenalidomide orally once a day. Lenalidomide dose was escalated by 5 mg in a step-wise manner every 28 days up to a maximum dose of 25 mg daily based on tolerability.
  Participants continued receiving study drug until disease progression or unacceptable toxicity, unless they withdrew consent or had other reasons to discontinue from study drug
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — Depending on the starting dose, subjects will be allocated in a double-blind fashion to three different regimens and will escalate every 28 days, based on individual subject tolerability, as follows:
  * Treatment Arm 1: 5 mg →10 mg →15 mg →20 mg →25 mg/daily
  * Treatment Arm 2: 10 mg →15 mg →20 mg →25 mg/daily
  * Treatment Arm 3: 15 mg →20 mg →25 mg/daily Subjects will continue treatment until disease progression or unacceptable toxicity

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of different dose regimens of lenalidomide in patients with relapsed or refractory chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of signing the informed consent form
* Must be able to adhere to the study visit schedule and other protocol requirements
* Must have a documented diagnosis of B-cell CLL
* Must be relapsed or refractory to at least 1 regimen for treatment of CLL. At least one of the prior treatments must have included a purine analog-based or bendamustine-based regimen
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Active infections requiring systemic antibiotics
* Systemic treatment for B-cell CLL within 28 days of initiation of lenalidomide treatment
* Alemtuzumab therapy within 120 days of initiating lenalidomide treatment
* Prior therapy with lenalidomide
* History of grade 4 rash due to prior thalidomide treatment
* Planned autologous or allogeneic bone marrow transplantation
* Central nervous system (CNS) involvement as documented by spinal fluid cytology or imaging.
* Uncontrolled hyperthyroidism or hypothyroidism
* Venous thromboembolism within 12 months
* ≥ Grade 2 neuropathy
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia
* Disease transformation [i.e. Richter's Syndrome (lymphomas) or prolymphocytic leukemia]
* Participation in any clinical study or having taken any investigational therapy within 28 days prior to initiating lenalidomide therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-10-19 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Jones, M.D., MPH, Study Director — Celgene Corporation
Locations (52):
- United States (16):
  - UCSD Moores Cancer Center, La Jolla, California
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - Stanford University School of Medicine, Stanford, California
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Cancer and Blood Disease Center, Lecanto, Florida
  - Northwestern University Medical Center Division of Hematology Oncology, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Karmanos Cancer Institute, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Long Island Jewish Medical Center CLL Research and Treatment Program, New Hyde Park, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Drexel University, College of Medicine, Clinical Research Group, Philadelphia, Pennsylvania
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
- France (14):
  - CHU Sud, Amiens
  - Hopital Avicenne, Bobigny
  - CHU Grenoble, Grenoble
  - Clinique Victor Hugo, Le Mans
  - Institut Paoli Calmettes, Marseille
  - CHU Montpellier - Hôpital Saint Eloi, Montpellier
  - Hopital Emile Muller, Mulhouse
  - Hopital Pitie Salpetriere, Paris
  - CH Perpignan - Hopital Saint-Jean, Perpignan
  - CHRU - Hopital du Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Robert Debre, Reims
  - CHU Rennes Hematology, Rennes
  - CHRU Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (6):
  - Charite -Universitätsmedizin Berlin, Berlin
  - Klinikum der Universitat zu Koln, Cologne
  - Universitatsklinikum Essen, Essen
  - Ernst-Moritz-Arndt-Universität Greifswald, Greifswald
  - Universitatsklinikum Schleswig Holstein, Kiel
  - University of Ulm Abteilung Innere Medizin III, Ulm
- Italy (6):
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Ematologia ed Immunologia, Azienda Ospedaliera "Vito Fazzi" di Lecce, Lecce
  - I.R.C.C.S. Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia - IEO, Milan
  - Universita degli Studi di Padova, Padua
  - Universita' Degli Studi Di Perugia, Perugia
- Spain (2):
  - Hospital Clinic Provincial de Barcelona, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
- Karolinska Universitetssjukhuset, Stockholm, Sweden
- United Kingdom (5):
  - St James's Institute of Oncology, Leeds
  - St.Bartholomew's Hospital, London
  - King's College Hospital, London
  - The Royal Marsden Hospital, London
  - Christie Hospital NHS Foundation Trust, Manchester

REFERENCES:
- [Background] Wendtner CM, Hallek M, Fraser GA, Michallet AS, Hillmen P, Durig J, Kalaycio M, Gribben JG, Stilgenbauer S, Buhler A, Kipps TJ, Purse B, Zhang J, De Bedout S, Mei J, Chanan-Khan A. Safety and efficacy of different lenalidomide starting doses in patients with relapsed or refractory chronic lymphocytic leukemia: results of an international multicenter double-blinded randomized phase II trial. Leuk Lymphoma. 2016;57(6):1291-9. doi: 10.3109/10428194.2015.1128540. Epub 2016 Jan 14. PMID 26763349
- [Background] Buhler A, Wendtner CM, Kipps TJ, Rassenti L, Fraser GA, Michallet AS, Hillmen P, Durig J, Gregory SA, Kalaycio M, Aurran-Schleinitz T, Trentin L, Gribben JG, Chanan-Khan A, Purse B, Zhang J, De Bedout S, Mei J, Hallek M, Stilgenbauer S. Lenalidomide treatment and prognostic markers in relapsed or refractory chronic lymphocytic leukemia: data from the prospective, multicenter phase-II CLL-009 trial. Blood Cancer J. 2016 Mar 11;6(3):e404. doi: 10.1038/bcj.2016.9. PMID 26967821

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 29 sites from North America and Europe.
Pre-assignment Details: Participants were randomized (1:1:1) in a double-blind fashion, according to age (< 65 versus ≥ 65 years) and disease status (relapsed versus refractory) to their last purine-analog or bendamustine-based prior regimen.
Period: Overall Study
Arm/Group | Lenalidomide 5 mg | Lenalidomide 10 mg | Lenalidomide 15 mg
Started | 34 | 35 | 35
Received Treatment | 34 | 34 | 35
Completed (completed represents participants who discontinued the study.) | 34 | 35 | 35
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lenalidomide 5 mg: Participants received a starting dose of 5 mg lenalidomide orally once a day. Lenalidomide dose was escalated by 5 mg in a step-wise manner every 28 days up to a maximum dose of 25 mg daily based on tolerability.
- Lenalidomide 10 mg: Participants received a starting dose of 10 mg lenalidomide orally once a day. Lenalidomide dose was escalated by 5 mg in a step-wise manner every 28 days up to a maximum dose of 25 mg daily based on tolerability.
- Lenalidomide 15 mg: Participants received a starting dose of 15 mg lenalidomide orally once a day. Lenalidomide dose was escalated by 5 mg in a step-wise manner every 28 days up to a maximum dose of 25 mg daily based on tolerability.
- Total: Total of all reporting groups
Arm/Group | Lenalidomide 5 mg | Lenalidomide 10 mg | Lenalidomide 15 mg | Total
Number analyzed (Participants) | 34 | 35 | 35 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.46) | 63.3 (8.31) | 63.7 (7.56) | 63.6 (8.39)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 16 | 19 | 17 | 52
  ≥ 65 years | 18 | 16 | 18 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 11 | 32
  Male | 26 | 22 | 24 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31 | 30 | 33 | 94
  Black or African American | 2 | 4 | 2 | 8
  Other | 0 | 1 | 0 | 1
  Unknown | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Adverse events (AEs) were graded for severity by the investigator according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0 with the exceptions of hematologic toxicities and tumor lysis syndrome, according to the following scale: Grade 1 = Mild Grade 2 = Moderate Grade 3 = Severe Grade 4 = Life Threatening or disabling AE Grade 5 = Death The investigator determined the relationship of each AE to study drug based on the timing of the AE and whether other medications, therapeutic interventions, or underlying conditions could provide a sufficient explanation for the observed event.
Time Frame: From first dose of study drug to 30 days after the last dose; the maximum duration of treatment was 251, 265, and 267 weeks in the 5 mg, 10 mg, and 15 mg treatment groups respectively.
Population: Randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide 5 mg | Lenalidomide 10 mg | Lenalidomide 15 mg
Number analyzed (Participants) | 34 | 34 | 35
Participants
  Any adverse events | 34 | 34 | 35
  Treatment-related adverse events (TRAE) | 33 | 34 | 32
  Grade 3/4 adverse events | 33 | 32 | 34
  Treatment-related Grade 3/4 adverse events | 31 | 32 | 30
  Grade 5 adverse events | 4 | 4 | 3
  Treatment-related Grade 5 adverse events | 2 | 2 | 0
  Serious adverse events | 24 | 24 | 27
  Treatment-related serious adverse events | 15 | 13 | 20
  AE leading to discontinuation of study drug | 21 | 17 | 16
  TRAE leading to discontinuation of study drug | 16 | 14 | 13
  AE leading to study drug dose reduction only | 8 | 6 | 5
  AE leading to study drug dose interruption only | 25 | 24 | 25
  AE leading to study drug interruption & reduction | 18 | 26 | 19

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of patients with a complete response (CR), CR with incomplete bone marrow (BM) recovery (CRi) or partial response (PR) during treatment. Response was assessed according to the 2008 International Workshop on Chronic Lymphocytic Leukemia (iwCLL) guidelines. Per the guidelines, a CR required peripheral blood lymphocytes below 4 x 10^9/L, absence of lymphadenopathy, no hepatomegaly or splenomegaly, absence of disease and blood counts neutrophils >1.5 x 10^9/L, platelets >100 x 10^9/L, hemoglobin (hgb) >11g/dL) and BM at least normocellular for age. CRi = CR with incomplete BM recovery. PR = required at least 2 months from end of treatment, a ≥50% decrease in peripheral blood lymphocyte count from the pre-treatment value and either a ≥ 50% reduction in lymphadenopathy or ≥50% reduction of liver enlargement or ≥50% reduction of spleen enlargement plus neutrophils >1.5 x 10^9/ or ≥50% increase, platelets >100 x 10^9/L or ≥50% increase, hgb 11 g/dL.
Time Frame: Response was assessed after 3 cycles of therapy (Week 12) and every 4 weeks thereafter until disease progression. Maximum time on study was 91 months.
Population: All randomized participants (intent-to-treat population)
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide 5 mg | Lenalidomide 10 mg | Lenalidomide 15 mg
Number analyzed (Participants) | 34 | 35 | 35
percentage of participants | 47.1 | 37.1 | 40.0

3. Secondary Outcome: Kaplan-Meier Estimate of Duration of Response
Description: Duration of response (DOR) was defined as the time from the first visit where PR, CRi, or CR was documented to progressive disease (PD). Duration of response was censored at the last date that the participant was known to be progression-free for participants who had not progressed at the time of analysis or who withdrew consent or were lost to follow-up prior to documentation of progression.
Time Frame: as for outcome 2
Population: Randomized participants with an objective response (CR/CRi or PR)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide 5 mg | Lenalidomide 10 mg | Lenalidomide 15 mg
Number analyzed (Participants) | 16 | 13 | 14
weeks | 101.1 [60.6 to 239.3] | 35.1 [22.0 to NA] — Could not be calculated due to the low number of events | 88.8 [72.1 to 127.3]

4. Secondary Outcome: Time to Response
Description: Time to response (TTR) was calculated as the time from randomization to the first documented date of response (PR, CRi or CR) based on iwCLL guidelines for participants with an objective response during the treatment period.
Time Frame: as for outcome 2
Population: Randomized participants with an objective response (CR/CRi or PR)
Measure: Median (Full Range); unit: weeks
Arm/Group | Lenalidomide 5 mg | Lenalidomide 10 mg | Lenalidomide 15 mg
Number analyzed (Participants) | 16 | 13 | 14
weeks | 16.9 [12.1 to 74.1] | 12.6 [8.4 to 52.1] | 12.7 [12.0 to 147.3]

5. Secondary Outcome: Kaplan-Meier Estimate of Time to Progression
Description: Time to progression (TTP) was defined as the time from randomization to the first documented progression. For participants who did not progress during the study, TTP was censored at the last adequate response assessment showing evidence of no disease progression.
Time Frame: From randomization until the end of the study; maximum time on study was 91 months.
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide 5 mg | Lenalidomide 10 mg | Lenalidomide 15 mg
Number analyzed (Participants) | 34 | 35 | 35
weeks | 96.3 [20.6 to 251.3] | 47.6 [31.9 to 261.1] | 66.3 [20.1 to 89.3]

6. Secondary Outcome: Kaplan-Meier Estimate of Event-Free Survival
Description: Event-free survival (EFS) is the interval between the start of treatment to the first sign of disease progression, or treatment for relapse or death (whichever occurred first). If withdrawal of consent or loss to follow-up occurred before documented progression or death, then these observations were censored at the date when the last complete tumor assessments determined a lack of progression.
Time Frame: From randomization until the end of the study; maximum time on study was 91 months.
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide 5 mg | Lenalidomide 10 mg | Lenalidomide 15 mg
Number analyzed (Participants) | 34 | 35 | 35
weeks | 25.6 [16.1 to 77.6] | 31.9 [21.1 to 47.6] | 24.1 [13.4 to 66.3]

7. Secondary Outcome: Kaplan-Meier Estimate of Progression Free Survival
Description: Progression-free survival (PFS) was calculated as the time from randomization to the first documented progression or death due to any cause during or after the treatment period, whichever occurred first. The progression date was assigned to the earliest time when any progression is observed without prior missing assessments. If withdrawal of consent or loss to follow-up occurred before documented progression or death, then these observations were censored at the date when the last complete tumor assessments determined a lack of progression.
Time Frame: From randomization until the end of the study; maximum time on study was 91 months.
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide 5 mg | Lenalidomide 10 mg | Lenalidomide 15 mg
Number analyzed (Participants) | 34 | 35 | 35
weeks | 31.4 [16.1 to 96.3] | 45.1 [22.4 to 120.1] | 66.3 [16.1 to 89.3]

8. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival
Description: Overall survival (OS) was defined as the time from randomization to death from any cause. Overall survival was censored at the last date that the participant was known to be alive for participants who were alive at the time of analysis and for participants who had withdrawn consent or were lost to follow-up before death was documented.
Time Frame: From randomization until the end of the study; maximum time on study was 91 months.
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide 5 mg | Lenalidomide 10 mg | Lenalidomide 15 mg
Number analyzed (Participants) | 34 | 35 | 35
weeks | 161.0 [64.9 to 209.0] | 106.7 [83.4 to 235.7] | 154.6 [80.9 to 214.7]

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after the last dose; the maximum duration of treatment was 251, 265, and 267 weeks in the 5 mg, 10 mg, and 15 mg treatment groups respectively.
Arm/Group | Lenalidomide 5 mg | Lenalidomide 10 mg | Lenalidomide 15 mg
All-Cause Mortality (participants affected / at risk) | 24/34 | 23/34 | 26/35
Serious Adverse Events (participants affected / at risk) | 24/34 | 24/34 | 27/35
Other Adverse Events (participants affected / at risk) | 34/34 | 34/34 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide 5 mg (N=34) | Lenalidomide 10 mg (N=34) | Lenalidomide 15 mg (N=35)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 4 | 4
IMMUNE THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 | 1 | 0
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 2 | 3
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 1 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 2
ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1
CARDIAC TAMPONADE (Cardiac disorders) | 0 | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 3 | 0
COLITIS (Gastrointestinal disorders) | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 1 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 0 | 1 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1
ASTHENIA (General disorders) | 0 | 0 | 1
DEATH (General disorders) | 1 | 0 | 0
DISEASE PROGRESSION (General disorders) | 0 | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 1 | 1
IMPAIRED HEALING (General disorders) | 0 | 1 | 0
PAIN (General disorders) | 0 | 0 | 1
PYREXIA (General disorders) | 2 | 1 | 2
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 1 | 0
ASPERGILLUS INFECTION (Infections and infestations) | 0 | 1 | 0
ATYPICAL PNEUMONIA (Infections and infestations) | 0 | 1 | 0
BACTERAEMIA (Infections and infestations) | 2 | 0 | 0
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 | 1 | 1
CELLULITIS (Infections and infestations) | 1 | 0 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0 | 1
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 | 0 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 1 | 0
EPIDIDYMITIS (Infections and infestations) | 0 | 1 | 0
EPIGLOTTITIS (Infections and infestations) | 0 | 0 | 1
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 0 | 0 | 1
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 1 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 1
GASTROENTERITIS SALMONELLA (Infections and infestations) | 0 | 0 | 1
HERPES ZOSTER (Infections and infestations) | 1 | 0 | 0
INFECTIOUS MONONUCLEOSIS (Infections and infestations) | 1 | 0 | 0
LUNG INFECTION (Infections and infestations) | 0 | 1 | 0
NEUTROPENIC INFECTION (Infections and infestations) | 1 | 1 | 0
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 1 | 0 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 1 | 0
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 | 2 | 0
PNEUMONIA (Infections and infestations) | 5 | 4 | 10
PNEUMONIA INFLUENZAL (Infections and infestations) | 1 | 1 | 0
POST PROCEDURAL CELLULITIS (Infections and infestations) | 0 | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1 | 2
SALMONELLOSIS (Infections and infestations) | 0 | 1 | 0
SEPSIS (Infections and infestations) | 1 | 1 | 1
SEPTIC SHOCK (Infections and infestations) | 0 | 0 | 1
SOFT TISSUE INFECTION (Infections and infestations) | 0 | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 0 | 1
SYSTEMIC MYCOSIS (Infections and infestations) | 0 | 1 | 0
TUBERCULOSIS OF PERIPHERAL LYMPH NODES (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 1
WOUND INFECTION (Infections and infestations) | 0 | 0 | 1
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 3 | 0 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 | 0 | 2
ARTHRITIS REACTIVE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
COCCYDYNIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
ACUTE LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
ANAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
MENINGIOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
NEUROFIBROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OLIGOASTROCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 6
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 1 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 0 | 2
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 2 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | 1 | 0 | 2
VENOUS THROMBOSIS LIMB (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide 5 mg (N=34) | Lenalidomide 10 mg (N=34) | Lenalidomide 15 mg (N=35)
ANAEMIA (Blood and lymphatic system disorders) | 11 | 18 | 15
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 2 | 0 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 2 | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 2
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 1 | 2 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 25 | 30 | 26
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 17 | 25 | 21
ANGINA PECTORIS (Cardiac disorders) | 0 | 1 | 2
TACHYCARDIA (Cardiac disorders) | 0 | 2 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 2
DRY EYE (Eye disorders) | 3 | 0 | 0
LACRIMATION INCREASED (Eye disorders) | 1 | 1 | 2
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 3 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 10 | 6
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 3 | 3
CONSTIPATION (Gastrointestinal disorders) | 11 | 13 | 13
DIARRHOEA (Gastrointestinal disorders) | 14 | 18 | 16
DRY MOUTH (Gastrointestinal disorders) | 1 | 2 | 6
DYSPEPSIA (Gastrointestinal disorders) | 1 | 3 | 0
DYSPHAGIA (Gastrointestinal disorders) | 3 | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 2 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 2 | 0
NAUSEA (Gastrointestinal disorders) | 10 | 15 | 11
ORAL PAIN (Gastrointestinal disorders) | 2 | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 3 | 1 | 4
VOMITING (Gastrointestinal disorders) | 8 | 5 | 8
ASTHENIA (General disorders) | 4 | 4 | 4
CHEST DISCOMFORT (General disorders) | 2 | 0 | 0
CHILLS (General disorders) | 0 | 2 | 6
FATIGUE (General disorders) | 18 | 17 | 23
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 3 | 0
LOCAL SWELLING (General disorders) | 1 | 2 | 0
MALAISE (General disorders) | 2 | 1 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 2 | 1
OEDEMA PERIPHERAL (General disorders) | 6 | 8 | 5
PYREXIA (General disorders) | 12 | 15 | 16
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 2
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 4 | 2 | 3
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 5 | 0 | 0
BRONCHITIS (Infections and infestations) | 5 | 2 | 3
CELLULITIS (Infections and infestations) | 0 | 2 | 2
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 2 | 0 | 0
HERPES SIMPLEX (Infections and infestations) | 0 | 0 | 4
LABYRINTHITIS (Infections and infestations) | 0 | 0 | 2
LOCALISED INFECTION (Infections and infestations) | 0 | 1 | 2
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 3 | 0 | 1
ORAL CANDIDIASIS (Infections and infestations) | 0 | 3 | 3
ORAL HERPES (Infections and infestations) | 2 | 3 | 4
OTITIS MEDIA (Infections and infestations) | 0 | 2 | 0
PHARYNGITIS (Infections and infestations) | 1 | 1 | 3
PNEUMONIA (Infections and infestations) | 2 | 4 | 5
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0
RHINITIS (Infections and infestations) | 1 | 3 | 2
SALMONELLOSIS (Infections and infestations) | 0 | 2 | 0
SINUSITIS (Infections and infestations) | 4 | 1 | 3
SKIN INFECTION (Infections and infestations) | 1 | 0 | 3
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 2 | 1
TOOTH INFECTION (Infections and infestations) | 1 | 0 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 | 5 | 3
URINARY TRACT INFECTION (Infections and infestations) | 4 | 5 | 2
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1 | 7
CONTUSION (Injury, poisoning and procedural complications) | 3 | 2 | 2
LACERATION (Injury, poisoning and procedural complications) | 2 | 0 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 2 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 6 | 7 | 5
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 4 | 5
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 | 3 | 1
BLOOD CREATININE INCREASED (Investigations) | 2 | 1 | 2
BLOOD IMMUNOGLOBULIN G DECREASED (Investigations) | 0 | 0 | 2
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 | 2 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 | 2 | 0
WEIGHT DECREASED (Investigations) | 7 | 13 | 10
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 | 11 | 9
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 2
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 2 | 2 | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 2 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 1
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 3 | 2 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 5 | 5 | 5
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 4 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 2
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 | 3 | 2
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 | 0 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 | 4 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 2 | 10
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 6 | 7 | 11
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 | 5 | 5
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 | 21 | 23
DIZZINESS (Nervous system disorders) | 6 | 1 | 4
DYSGEUSIA (Nervous system disorders) | 3 | 0 | 3
HEADACHE (Nervous system disorders) | 5 | 4 | 4
HYPOAESTHESIA (Nervous system disorders) | 2 | 2 | 2
LETHARGY (Nervous system disorders) | 2 | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 3 | 1 | 2
PARAESTHESIA (Nervous system disorders) | 2 | 2 | 3
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 | 0 | 2
SOMNOLENCE (Nervous system disorders) | 1 | 2 | 0
TREMOR (Nervous system disorders) | 2 | 2 | 0
ANXIETY (Psychiatric disorders) | 0 | 1 | 4
DEPRESSION (Psychiatric disorders) | 1 | 3 | 2
INSOMNIA (Psychiatric disorders) | 3 | 4 | 8
DYSURIA (Renal and urinary disorders) | 2 | 4 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 2 | 1
POLLAKIURIA (Renal and urinary disorders) | 2 | 1 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 | 15 | 12
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 9
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 9
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 5 | 1
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 2 | 7
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 6 | 10 | 11
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 4 | 3
RASH (Skin and subcutaneous tissue disorders) | 9 | 8 | 16
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
RASH MACULAR (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
URTICARIA PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
HYPOTENSION (Vascular disorders) | 4 | 4 | 5
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Study Protocol (2015-04-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT00963105/Prot_000.pdf
  • Statistical Analysis Plan (2012-11-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT00963105/SAP_001.pdf